CLINICAL TRIAL: NCT01783509
Title: Longitudinal Assessment and Genetic Understanding of Limb-Girdle Muscular Dystrophy
Brief Title: Limb Girdle Muscular Dystrophy (LGMD) Natural History
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Sponsor
Other Study IDs: LGMD Nat Hx
Record Dates: First submitted 2013-01-18; First posted 2013-02-05 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2017-07

CONDITIONS: Muscular Dystrophies, Limb-Girdle (GENETICALLY CONFIRMED)
Keywords: GENETICALLY CONFIRMED limb girdle muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LGMD: Patients with GENETICALLY CONFIRMED limb girdle muscular dystrophy

SUMMARY:
The purpose of this study is to understand more about limb-girdle muscular dystrophy. Therefore, the investigators would like to track the following information collected once a year from patients with GENETICALLY CONFIRMED LGMD: quality of life questionnaires, muscle strength, motor function, routine examination, assessment of patient (or parent) understanding of LGMD, and serum (blood) for growth factors, cytokines, and biomarkers (all parts of your blood). By tracking this information, we hope to be able to understand more about the diagnosis, progression and natural history of this disorder.

ELIGIBILITY:
Inclusion Criteria:

* You have a GENETICALLY CONFIRMED diagnosis of Limb Girdle Muscular Dystrophy
* You must be at least 6 years of age or older (if under 18 you will need Parental consent)
* You must be able to travel to the study site
* You must be able to provide a DNA/Gene testing report that confirms a diagnosis of LGMD

Exclusion Criteria:

* You or your child do not have a diagnosis of LGMD
* Your child is under age 6
* You or your child are not able to travel to the study site

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of GENETICALLY CONFIRMED LGMD
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Comprehensive clinical evaluation of individuals with GENETICALLY CONFIRMED LGMD, according to the study protocol, in order to evaluate disease progression | yearly up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Binalsheikh, MD, Principal Investigator — Carolinas Medical Center - Pediatrics
Locations (1):
- Carolinas Medical Center - Pediatrics, Charlotte, North Carolina, United States